CLINICAL TRIAL: NCT03344120
Title: Comparison Between Symptomps Related to Pigtail Suture Stent Versus Conventional Double J After Ureterorenoscopy for Stone Treatment. A Prospective Randomized Trial
Brief Title: Symptoms Comparison: Suture-stent vs Conventional Double-J Stents After Ureterorenoscopy. A Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Andrea Bosio, MD Urologist, PhD, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOUCSSTURAB004
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Symptoms and Signs; Pain; Ureteral Calculi
Keywords: Symptoms and Signs; Pain; Ureteral Calculi; Ureteroscopy; Ureteral Stents
MeSH Terms: conditions — Signs and Symptoms; Pain; Ureteral Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suture stent (Active Comparator): suture stent positioning after ureteroscopy. Intervention: administration of USSQ questionnaire.
  Interventions: Other: Administration of USSQ Symptoms questionnaire after stent positioning
- conventional double-J stent (Active Comparator): conventional double-J stent positioning after ureteroscopy. Intervention: administration of USSQ questionnaire.
  Interventions: Other: Administration of USSQ Symptoms questionnaire after stent positioning

INTERVENTIONS:
Other: Administration of USSQ Symptoms questionnaire after stent positioning — Administration of USSQ Symptoms questionnaire to patients with two different type of stents after ureteroscopy

SUMMARY:
Double J ureteral stents (DJ) are widely used in urological practice and commonly inserted after most of ureteroscopies. Stent-related symptoms (SRS) represent a major issue. Many research lines have been explored with the aim of decreasing SRS: Vogt et al. projected a self-made pigtail suture stent (PSS) replacing the distal pigtail with a 0.3 Fr suture reaching the bladder, showing decreased SRS and good tolerance. To date, these promising results hasn't been confirmed by a prospective randomized controlled trial (RCT) involving a marketed PSS. Thus, we designed a prospective single-blind RCT to compare SRS caused by marketed PSS and conventional DJ after uncomplicated URS for stone treatment.

ELIGIBILITY:
Inclusion Criteria:

* ureteral or renal stones < 2 cm needing treatment through semirigid or flexible URS and laser lithotripsy
* stone-free procedure and absence of intraprocedural complications
* WHO performance status 0-2

Exclusion Criteria:

* significant residual fragments at the end of the procedure
* intraprocedural complications (e.g. ureteral damage or stricture)
* indwelling double J stent
* acute kidney failure
* urinary tract infection
* urinary tract abnormalities
* pathologies or medications potentially influencing voiding pattern and pain perception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Urinary Symptom Index Score | 14 days
  to compare Urinary Symptom Index Score (sum of USSQ Urinary symptoms scores) of suture stent and double J group, 2 weeks after surgery.

SECONDARY OUTCOMES:
USSQ domains' scores | 14 days
  to compare USSQ domains' scores of suture stent and double J group, 2 weeks after surgery
USSQ domains' scores | 2 days
  to compare USSQ domains' scores of suture stent and double J group, 2 days after surgery
USSQ single answers | 14 day
  to compare USSQ single answers of suture stent and double J group, 2 weeks after surgery
USSQ single answers | 2 days
  to compare USSQ single answers of suture stent and double J group, 2 days after surgery
2 weeks USSQ domains' subscores adjusted for baseline | 6 weeks
  to compare 2 weeks USSQ domains' subscores adjusted for baseline of suture stent and double J group
complications and adverse events | 2 weeks
  to compare complications and adverse events of suture stent and double J group

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bosio, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosio A, Alessandria E, Agosti S, Vitiello F, Vercelli E, Bisconti A, Piana P, Fop F, Gontero P. Pigtail Suture Stents Significantly Reduce Stent-related Symptoms Compared to Conventional Double J Stents: A Prospective Randomized Trial. Eur Urol Open Sci. 2021 May 10;29:1-9. doi: 10.1016/j.euros.2021.03.011. eCollection 2021 Jul. PMID 34337527